CLINICAL TRIAL: NCT02329093
Title: Non-weight Bearing in Hip Joint With Accompanying Joint Pain Might Not Progress Radiographic OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Assistant Professor, Shinshu University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hip OA Pro-Study 2015
Record Dates: First submitted 2014-12-21; First posted 2014-12-31 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Hip OA
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone Signal Changes (Experimental)
  Interventions: Procedure: To MRI-detecting bone signal changes in radiographic hip OA

INTERVENTIONS:
Procedure: To MRI-detecting bone signal changes in radiographic hip OA — To examine whether or not non-weight bearing reduced OA progression

SUMMARY:
As we have previously reported, the primary cause of hip OA with accompanying joint pain might be bone alterations which can be microfracture. In order to prove it, it is planned that conservative treatment will be performed on the hip OA patients with accompanying joint pain for the first year. For the second year, if the patients still have joint pain, they will do non-weght bearing walk.

ELIGIBILITY:
Inclusion Criteria:

* Hip OA, Joint pain

Exclusion Criteria:

* Obvious radipgraphic fracture in hip joint,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Bone Signal Changes on the Hip MRI | 1 - 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan